CLINICAL TRIAL: NCT05692453
Title: Pulse Oximetry Accuracy by Skin Color
Status: Not yet recruiting | Type: Observational
Sponsor: Brittany Willer (Other)
Responsible Party: Sponsor-Investigator, Brittany Willer, Director of Quality Improvement & Safety, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: STUDY00003117
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Surgery
MeSH Terms: interventions — Blood Gas Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Diagnostic Test: Arterial blood gas with co-oximetry — 1 mL blood sample for ABG-CoOx analysis to obtain co-oximetry measured arterial oxygen saturation (SaO2C) and standard ABG derived arterial oxygen saturation (SaO2S).
  Other Names: ABG-CoOx

SUMMARY:
This is a prospective, non-randomized, non-blinded comparative study to evaluate the accuracy of pulse oximetry compared to co-oximetry in dark-skinned (Black) compared to lighter-skinned (White) children undergoing anesthesia, using standard FDA performance statistics as measured by mean bias and accuracy root mean squared to evaluate device performance.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, non-blinded comparative study.

There will be no changes to the anesthetic or surgical plan to accommodate this study. Patients undergoing anesthesia will be induced per their anesthetic team. Following endotracheal intubation, the patient will be placed on air (FiO2 21%) at 4 liters per minute fresh gas flow. After a minimum of 3 minutes has elapsed, the anesthesia team will obtain an arterial blood sample of approximately 1 mL. This can be obtained from an arterial line if one is planned for the procedure or already in place by accessing the line per standard procedure. If an arterial line is not placed, the arterial sample will be obtained by percutaneous arterial puncture using ultrasound guidance and a 25-gauge blood gas syringe. The patient's SpO2 will be noted using a pulse oximetry probe placed on the right index finger when the arterial sample is drawn, along with the date/time of sample acquisition. Once the sample is drawn, the patient's anesthetic and surgery will proceed as per his anesthesia team. The arterial sample will be immediately delivered to the Nationwide Children's Hospital laboratory for simultaneous ABG and ABG-CoOx analysis to obtain SaO2S and SaO2C, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-9 years undergoing general anesthesia with or without arterial line placement.

Exclusion Criteria:

* Patients with cyanotic congenital heart disease.
* Patients with bleeding disorders.
* Patients taking blood thinners.

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children undergoing surgery at Nationwide Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Pulse Oximetry | Baseline
  Accuracy of pulse oximetry readings (SpO2) as compared with arterial oxygen saturations measured by arterial blood gas with co-oximetry (ABG-CoOx).

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Willer, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No